CLINICAL TRIAL: NCT00308139
Title: A Randomized, Open-Label, Multicenter, Comparator-Controlled Study to Examine the Effects of Exenatide Long-Acting Release on Glucose Control (HbA1c) and Safety in Subjects With Type 2 Diabetes Mellitus Managed With Diet Modification and Exercise and/or Oral Antidiabetic Medications
Brief Title: Effects of Exenatide Long-Acting Release on Glucose Control and Safety in Subjects With Type 2 Diabetes Mellitus(DURATION - 1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2993LAR-105 (DURATION - 1); MB001-010 (Other: Bristol Myers Squibb)
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Results first posted 2012-08-17 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide; long acting release; LAR; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide Once Weekly (Experimental): Subcutaneous injection (SC), once a week of long acting release (LAR) exenatide.
  Interventions: Drug: exenatide, long acting release
- Exenatide Twice Daily (Active Comparator): subcutaneous injection (SC), twice a day for the first 30 weeks, followed by exenatide LAR SC injection weekly for the remainder of the study.
  Sub-study: Exenatide 2 mg subcutaneous injection, Administered Using the Exenatide Once Weekly Single-Dose Tray , once a week for 11 visits, switch to Exenatide 2 mg subcutaneous injection, Administered Using the Dual chamber pen device. Exenatide 2mg SC injection administered using the Dual chamber pen device.
  Interventions: Drug: exenatide

INTERVENTIONS:
Drug: exenatide, long acting release
  Other Names: BYDUREON
  Arms: Exenatide Once Weekly
Drug: exenatide
  Other Names: Byetta
  Arms: Exenatide Twice Daily

SUMMARY:
A Randomized, Open-Label, Multicenter, Comparator-Controlled Study to Examine the Effects of Exenatide Long-Acting Release (LAR) on Glucose Control (HbA1c) and Safety in Subjects with Type 2 Diabetes Mellitus Managed with Diet Modification and Exercise and/or Oral Antidiabetic Medications.

DETAILED DESCRIPTION:
This trial is designed to examine the effect of exenatide once weekly compared to exenatide twice daily on glucose control and safety in subjects for at least 30 weeks. The study is also designed to examine glucose control during the transition from exenatide twice daily for 30 weeks to exenatide once weekly. Long-term safety and efficacy will be monitored during the open-ended assessment periods. This study will be conducted in approximately 300 subjects with type 2 diabetes treated with diet modification and exercise alone or in combination with a stable regimen of metformin, SU, thiazolidinedione (TZD), a combination of metformin and SU, a combination of metformin and TZD, or a combination of SU and TZD.

ELIGIBILITY:
Inclusion Criteria:

* Has type 2 diabetes mellitus treated with diet modification and exercise alone or in combination with a stable regimen of a combination of metformin, sulphonylureas, and thiazolidinediones for a minimum of 2 months at screening.
* Hemoglobin A1c (HbA1c) of 7.1% to 11.0%, inclusive, at screening.
* Body mass index (BMI) of 25 kg/m2 to 45 kg/m2, inclusive, at screening.
* (For sub-study) Currently participating in open ended assessment period of main study 2993 LAR105

Exclusion Criteria:

* Has been previously exposed to exenatide (Byetta®), exenatide LAR, or any glucagon-like peptide-1 (GLP-1) analog.
* Received any investigational drug or has participated in any type of clinical trial within 30 days prior to screening.
* Has been treated, is currently treated, or is expected to require or undergo treatment with any of the following excluded medications:

  * Alpha glucosidase inhibitor or meglitinide within 30 days of screening;
  * Insulin within 2 weeks prior to screening or insulin for longer than 1 week within 3 months of screening;
  * Regular use (> 14 days) of drugs that directly affect gastrointestinal motility;
  * Regular use (> 14 days) of systemic corticosteroids by oral, intravenous, or intramuscular route; or potent, inhaled, or intrapulmonary steroids known to have a high rate of systemic absorption;
  * Regular use (> 14 days) of medications with addictive potential such as opiates and opioids;
  * Prescription or over-the-counter weight loss medications within 6 months of screening.
* (For sub-study) Subjects will be terminated from study who do not participate in the dual chamber pen substudy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2006-04; Primary Completion 2008-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Porter, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (25):
- United States (24):
  - Research Site 182, Encino, California
  - Research Site 171, La Jolla, California
  - Research Site 518, San Diego, California
  - Research Site 024, Walnut Creek, California
  - Research Site, Colorado Springs, Colorado
  - Research Site 057, Miami, Florida
  - Research Site, Chicago, Illinois
  - Research Site 149, Indianapolis, Indiana
  - Research Site 099, Lexington, Kentucky
  - Research Site 017, Detroit, Michigan
  - Research Site 224, Minneapolis, Minnesota
  - Research Site 312, St Louis, Missouri
  - Research Site 023, Butte, Montana
  - Research Site 053, Rochester, New York
  - Research Site 002, Durham, North Carolina
  - Research Site 123, Winston-Salem, North Carolina
  - Research Site 405, Cincinnati, Ohio
  - Research Site 557, Marion, Ohio
  - Research Site 231, Portland, Oregon
  - Research Site 152, Philadelphia, Pennsylvania
  - Research Site 587, Greer, South Carolina
  - Research Site 015, Dallas, Texas
  - Research Site 009, San Antonio, Texas
  - Research Site 108, Olympia, Washington
- Research Site, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Philis-Tsimikas A, Wysham CH, Hardy E, Han J, Iqbal N. Efficacy and tolerability of exenatide once weekly over 7 years in patients with type 2 diabetes: An open-label extension of the DURATION-1 study. J Diabetes Complications. 2019 Mar;33(3):223-230. doi: 10.1016/j.jdiacomp.2018.11.012. Epub 2018 Dec 5. PMID 30600137
- [Derived] Henry RR, Klein EJ, Han J, Iqbal N. Efficacy and Tolerability of Exenatide Once Weekly Over 6 Years in Patients with Type 2 Diabetes: An Uncontrolled Open-Label Extension of the DURATION-1 Study. Diabetes Technol Ther. 2016 Nov;18(11):677-686. doi: 10.1089/dia.2016.0107. Epub 2016 Aug 15. PMID 27525540
- [Derived] Wysham CH, MacConell LA, Maggs DG, Zhou M, Griffin PS, Trautmann ME. Five-year efficacy and safety data of exenatide once weekly: long-term results from the DURATION-1 randomized clinical trial. Mayo Clin Proc. 2015 Mar;90(3):356-65. doi: 10.1016/j.mayocp.2015.01.008. PMID 25744115
- [Derived] Grimm M, Han J, Weaver C, Griffin P, Schulteis CT, Dong H, Malloy J. Efficacy, safety, and tolerability of exenatide once weekly in patients with type 2 diabetes mellitus: an integrated analysis of the DURATION trials. Postgrad Med. 2013 May;125(3):47-57. doi: 10.3810/pgm.2013.05.2660. PMID 23748506
- [Derived] Macconell L, Pencek R, Li Y, Maggs D, Porter L. Exenatide once weekly: sustained improvement in glycemic control and cardiometabolic measures through 3 years. Diabetes Metab Syndr Obes. 2013;6:31-41. doi: 10.2147/DMSO.S35801. Epub 2013 Jan 21. PMID 23358123
- [Derived] Chiquette E, Toth PP, Ramirez G, Cobble M, Chilton R. Treatment with exenatide once weekly or twice daily for 30 weeks is associated with changes in several cardiovascular risk markers. Vasc Health Risk Manag. 2012;8:621-9. doi: 10.2147/VHRM.S37969. Epub 2012 Nov 12. PMID 23166441
- [Derived] Fineman MS, Mace KF, Diamant M, Darsow T, Cirincione BB, Booker Porter TK, Kinninger LA, Trautmann ME. Clinical relevance of anti-exenatide antibodies: safety, efficacy and cross-reactivity with long-term treatment. Diabetes Obes Metab. 2012 Jun;14(6):546-54. doi: 10.1111/j.1463-1326.2012.01561.x. Epub 2012 Feb 10. PMID 22236356
- [Derived] Taylor K, Gurney K, Han J, Pencek R, Walsh B, Trautmann M. Exenatide once weekly treatment maintained improvements in glycemic control and weight loss over 2 years. BMC Endocr Disord. 2011 Apr 29;11:9. doi: 10.1186/1472-6823-11-9. PMID 21529363
- [Derived] Buse JB, Drucker DJ, Taylor KL, Kim T, Walsh B, Hu H, Wilhelm K, Trautmann M, Shen LZ, Porter LE; DURATION-1 Study Group. DURATION-1: exenatide once weekly produces sustained glycemic control and weight loss over 52 weeks. Diabetes Care. 2010 Jun;33(6):1255-61. doi: 10.2337/dc09-1914. Epub 2010 Mar 9. PMID 20215461
- [Derived] Drucker DJ, Buse JB, Taylor K, Kendall DM, Trautmann M, Zhuang D, Porter L; DURATION-1 Study Group. Exenatide once weekly versus twice daily for the treatment of type 2 diabetes: a randomised, open-label, non-inferiority study. Lancet. 2008 Oct 4;372(9645):1240-50. doi: 10.1016/S0140-6736(08)61206-4. Epub 2008 Sep 7. PMID 18782641

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide Once Weekly -> Exenatide Once Weekly: Subcutaneous injection of 2 mg exenatide, once a week.
- Exenatide Twice Daily -> Exenatide Once Weekly: Subcutaneous injection of exenatide, twice a day (5 mcg exenatide per dose for first 4 weeks, then 10 mcg exenatide per dose for 26 weeks) followed by 2 mg exenatide, once a week.
Period: Overall Study
Arm/Group | Exenatide Once Weekly -> Exenatide Once Weekly | Exenatide Twice Daily -> Exenatide Once Weekly
Started | 152 | 151
Intent to Treat (ITT) | 148 (Subjects who received at least one injection of lead-in exenatide 5 mcg.) | 147 (Subjects who received at least one injection of lead-in exenatide 5 mcg.)
ITT in the 30-Week Assessment | 148 (ITT Subjects who received at least one injection of randomized dose.) | 145 (ITT Subjects who received at least one injection of randomized dose.)
Pharmacokinetics Population | 129 | 0
Evaluable Meal Tolerance Cohort | 27 | 24
30-Week Completed | 128 (Subjects who completed 30 weeks of assessment) | 130 (Subjects who completed 30 weeks of assessment)
Completed | 58 (Subjects who completed 364 weeks of assessment) | 64 (Subjects who completed 364 weeks of assessment)
Not Completed | 94 | 87
Not completed — Adverse Event | 20 | 14
Not completed — Lost to Follow-up | 13 | 8
Not completed — Protocol Violation | 3 | 2
Not completed — Withdrawal of Consent | 40 | 42
Not completed — Investigator Decision | 11 | 10
Not completed — Loss of Glucose Control | 5 | 7
Not completed — Administrative | 1 | 4
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Once Weekly -> Exenatide Once Weekly | Exenatide Twice Daily -> Exenatide Once Weekly | Total
Number analyzed (Participants) | 148 | 147 | 295
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 122 | 123 | 245
  >=65 years | 26 | 24 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (9.72) | 54.9 (9.63) | 55.0 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 72 | 138
  Male | 82 | 75 | 157
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of total hemoglobin] | 8.3 (0.99) | 8.3 (1.00) | 8.3 (0.99)
Weight [Mean (Standard Deviation); unit: kg] | 101.7 (18.76) | 101.9 (21.05) | 101.8 (19.90)
Background Oral Antidiabetic Agent [Number; unit: participants]
  Diet and Exercise | 21 | 22 | 43
  Metformin (MET) | 56 | 50 | 106
  Sulfonylurea (SU) | 6 | 10 | 16
  Thiazolidinediones (TZD) | 2 | 7 | 9
  MET+SU | 43 | 39 | 82
  MET+TZD | 14 | 14 | 28
  SU+TZD | 5 | 5 | 10
  SU+MET+TZD | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 30
Description: Absolute change in HbA1c from Baseline (Day -3) to Week 30 [Week 30 - Baseline]
Time Frame: Day -3, Week 30
Population: The ITT Population consisted of all randomized subjects who received at least one injection of study medication. Missing data up to Week 30 were imputed using the last observation carried forward (LOCF) approach for subjects who had data for at least one scheduled visit (including Early Termination) subsequent to the baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: percentage of total hemoglobin
Groups:
- Exenatide Once Weekly: Subcutaneous injection of 2 mg exenatide, once a week.
- Exenatide Twice Daily: Subcutaneous injection of exenatide, twice a day (5 mcg exenatide per dose for first 4 weeks, then 10 mcg exenatide per dose for 26 weeks) followed by 2 mg exenatide, once a week.
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 148 | 147
percentage of total hemoglobin | -1.87 (0.082) [-2.03 to -1.71] | -1.54 (0.082) [-1.70 to -1.38]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Superiority of exenatide long-acting release (LAR) once weekly to BYETTA if the upper limit of the 2-sided 95% confidence interval (CI) for treatment difference (LAR minus BYETTA) is less than 0; non-inferiority if this upper limit is less than 0.4%. Power:Assuming 20% dropout rate with 246 subjects will complete the study. This sample size would provide 90% power for non-inferiority test with assumption of greater reduction (0.1%) in LAR and a common standard deviation of 1.2%; Test type: Non-Inferiority or Equivalence — The choice of a 0.4% noninferiority margin was resulted from the considerations of expected clinical benefit of BYETTA in this study based on clinical data evaluating exenatide LAR and BYETTA, regulatory guidance, published literature, and statistical considerations; p = 0.0023, ANOVA; Analysis of variance (ANOVA) model includes treatment, baseline HbA1c stratum (<9% or >=9%), and concomitant SU use at screening as factors; Least Squares Mean Difference = -0.33, 95% CI 2-sided [-0.54 to -0.12], Standard Error of Mean 0.107

2. Secondary Outcome: Change in HbA1c From Baseline to Week 364
Description: Absolute change in HbA1c from Baseline (Day -3) to Week 364
Time Frame: Day -3, Week 364
Population: 7-Year Completer Population. Missing data up to Week 364 were imputed using the last observation carried forward (LOCF) approach for subjects who had data for at least one scheduled visit (including Early Termination) subsequent to the baseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of total hemoglobin
Arm/Group | Exenatide Once Weekly -> Exenatide Once Weekly | Exenatide Twice Daily -> Exenatide Once Weekly | All Treatment
Number analyzed (Participants) | 58 | 64 | 122
percentage of total hemoglobin | -1.49 (0.155) [-1.80 to -1.19] | -1.57 (0.144) [-1.85 to -1.28] | -1.53 (0.115) [-1.76 to -1.31]

3. Primary Outcome: Sub-study Relative Bioavailability of Exenatide When Administered Using the Exenatide Once Weekly Dual Chambered Pen and the Exenatide Once Weekly Single Dose Tray (Single Dose Tray-11 Weekly Doses Switch to Dual Chamber Pen-11 Weekly Dose)
Description: Measure by Geometric mean ratio (GMR) of plasma exenatide average steady state concentration Css,avg at Visit 11-14 to Visit 24-27 with 90% confidence interval
Time Frame: Week 22
Reporting Status: Not Posted

4. Secondary Outcome: Percentage of Subjects Achieving HbA1c Target of <7%
Description: Percentage of subjects achieving HbA1c target value of <7% at Week 30.
Time Frame: Week 30
Population: ITT Population. Missing data up to Week 30 were imputed using LOCF for subjects who had data for at least one scheduled visit (including Early Termination) subsequent to the baseline measurement. Subjects without post-baseline measurement were categorized as not achieving goal.
Measure: Number; unit: percentage of subjects
Groups:
- Exenatide Twice Daily: Subcutaneous injection of exenatide, twice a day (5 mcg exenatide per dose for first 4 weeks, then 10 mcg exenatide per dose for 26 weeks).
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 148 | 147
percentage of subjects | 70.9 | 51.0
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Analysis: Percentages of subjects achieving HbA1c target value of <7% at Week 30 were compared between treatments using a Cochran-Mantel-Haenszel (CMH) test, in which baseline HbA1c stratum (<9% or >=9%) and concomitant SU use at screening served as the stratification factors. Null hypothesis: no difference between treatments in percentage of subjects achieving HbA1c target. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.0003, Cochran-Mantel-Haenszel

5. Secondary Outcome: Percentage of Subjects Achieving HbA1c Target of <7%
Description: Percentages of subjects achieving HbA1c target value of <7% at Week 364
Time Frame: Week 364
Population: 7-Year Completer Population. Missing data up to Week 364 were imputed using LOCF for subjects who had data for at least one scheduled visit (including Early Termination) subsequent to the baseline measurement. Subjects without post-baseline measurement were categorized as not achieving goal.
Measure: Number; unit: percentage of subjects
Arm/Group | Exenatide Once Weekly -> Exenatide Once Weekly | Exenatide Twice Daily -> Exenatide Once Weekly | All Treatment
Number analyzed (Participants) | 58 | 64 | 122
percentage of subjects | 41.4 | 50.0 | 45.9

6. Secondary Outcome: Percentage of Subjects Achieving HbA1c Target of <=6.5%
Description: Percentages of subjects achieving HbA1c target values of <=6.5% at Week 30.
Time Frame: Week 30
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 148 | 147
percentage of subjects | 3.0 | 16.3
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Analysis: Percentage of subjects achieving HbA1c target value of <=6.5% at Week 30 were compared between treatments using CMH test, in which baseline HbA1c stratum (<9% or >=9%) and concomitant SU use at screening served as the stratification factors. Null hypothesis: no difference between treatments in percentage of subjects achieving HbA1c target. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.2042, Cochran-Mantel-Haenszel

7. Secondary Outcome: Percentage of Subjects Achieving HbA1c Target of <=6.5%
Description: Percentages of subjects achieving HbA1c target values of <=6.5% at Week 364
Time Frame: Week 364
Population: as for outcome 5
Measure: Number; unit: percentage of subjects
Arm/Group | Exenatide Once Weekly -> Exenatide Once Weekly | Exenatide Twice Daily -> Exenatide Once Weekly | All Treatmeat
Number analyzed (Participants) | 58 | 64 | 122
percentage of subjects | 22.4 | 37.5 | 30.3

8. Secondary Outcome: Percentage of Subjects Achieving HbA1c Target of <=6.0%
Description: Percentage of subjects achieving HbA1c target values of <=6.0% at Week 30.
Time Frame: Week 30
Population: as for outcome 4
Measure: Number; unit: percentage of subjects
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 148 | 147
percentage of subjects | 23.0 | 16.3
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Analysis: Percentages of subjects achieving HbA1c target values of <=6.0% at Week 30 were compared between treatments using CMH test, in which baseline HbA1c stratum (<9% or >=9%) and concomitant SU use at screening served as the stratification factors. Null hypothesis: no difference between treatments in percentage of subjects achieving HbA1c target. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.1513, Cochran-Mantel-Haenszel

9. Secondary Outcome: Exenatide LAR Steady State Concentration From Week 29 to Week 30
Description: Steady-state plasma exenatide concentration over the dosing interval of Week 29 to Week 30 (0-168 hours) was evaluated. Geometric mean for the average steady-state concentration and its 10th and 90th percentiles were reported.
Time Frame: Week 29 to Week 30
Population: The Pharmacokinetics Population consisted of subjects who received exenatide LAR treatment, and had adequate plasma exenatide concentration-time data to allow for reliable evaluation of exenatide LAR pharmacokinetics.
Measure: Geometric Mean (Inter-Quartile Range); unit: pg/mL
Arm/Group | Exenatide Once Weekly
Number analyzed (Participants) | 114
pg/mL | 300.23 [145.13 to 702.21]

10. Secondary Outcome: Change in 2 Hours (2h) Postprandial Glucose From Baseline to Week 14
Description: Change in 2h Postprandial Glucose from baseline (Day -3) to Week 14
Time Frame: Day -3, Week 14
Population: Evaluable Meal Tolerance Cohort consisted of ITT subjects who participated in the meal tolerance test and had adequate data to allow the reliable assessment of pharmacodynamics. Only subjects with non-missing baseline and Week 14 values were included in analysis.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 22 | 21
mg/dL | -95.88 (8.420) [-112.92 to -78.83] | -125.96 (8.292) [-142.74 to -109.17]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Analysis: Change in 2h postprandial glucose from baseline (Day -3) to Week 14 was analyzed using an ANCOVA model including treatment, baseline HbA1c stratum (<9% or >=9%), and concomitant SU use at screening as factors, and baseline value of the 2h postprandial glucose as a covariate. Null hypothesis: no difference between treatments in change from baseline 2h postprandial glucose; Test type: Superiority or Other; p = 0.0124, ANCOVA; Least Squares Mean Difference = 30.08, 95% CI 2-sided [6.88 to 53.28], Standard Error of Mean 11.458

11. Secondary Outcome: Sub-study Safety and Tolerability of Exenatide When Administered Using the Once Weekly Single Dose Tray and the Once Weekly Dual (Single Dose Tray-11 Weekly Doses Switch to Dual Chamber Pen-11 Weekly Dose)
Description: Measure by geometric mean ratio of the maximum steady state plasma exenatide concentration Css, max at Visit 11-14 to Visit 24-27 with 90% confidence interval and incidence of treatment-emergent injection site adverse events.
Time Frame: Week 22
Reporting Status: Not Posted

12. Secondary Outcome: Change in Body Weight From Baseline to Week 30
Description: Change in body weight from baseline (Day -3) to Week 30
Time Frame: Day -3, Week 30
Population: ITT Population. Missing data up to Week 30 were imputed using the LOCF approach for subjects who had data for at least one scheduled visit (including Early Termination) subsequent to the baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: kg
Groups:
- Exenatide Twice Daily: Subcutaneous injection of exenatide, twice a day (5 mcg exenatide per dose for first 4 weeks, then 10 mcg exenatide per dose for 26 week).
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 148 | 147
kg | -3.67 (0.468) [-4.59 to -2.75] | -3.59 (0.468) [-4.51 to -2.67]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Analysis: Change in body weight from baseline (Day -3) to Week 30 was analyzed using an analysis of covariance (ANCOVA) model including treatment, baseline HbA1c stratum (<9% or >=9%), and concomitant SU use at screening as factors, and baseline value of the body weight as a covariate. Null hypothesis: no difference between treatments in change from baseline body weight. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.8916, ANCOVA; Least Squares Mean Difference = -0.08, 95% CI 2-sided [-1.29 to 1.12], Standard Error of Mean 0.612

13. Secondary Outcome: Change in Body Weight From Baseline to Week 364
Description: Change in body weight from baseline (Day -3) to Week 364
Time Frame: Day -3, Week 364
Population: 7-Year Completer Population. Missing data up to Week 364 were imputed using the LOCF approach for subjects who had data for at least one scheduled visit (including Early Termination) subsequent to the baseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Arm/Group | Exenatide Once Weekly -> Exenatide Once Weekly | Exenatide Twice Daily -> Exenatide Once Weekly | All Treatment
Number analyzed (Participants) | 58 | 64 | 122
kg | -5.25 (0.468) [-7.23 to -3.27] | -2.71 (0.468) [-4.55 to -0.87] | -3.87 [-5.36 to -2.37]

14. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline to Week 30
Description: Change in fasting plasma glucose from baseline (Day -3) to Week 30.
Time Frame: Day -3, Week 30
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 148 | 147
mg/dL | -41.5 (2.97) [-47.4 to -35.7] | -24.6 (2.90) [-30.3 to -18.9]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Analysis: Change in fasting plasma glucose from baseline (Day -3) to Week 30 was analyzed using an ANCOVA model including treatment, baseline HbA1c stratum (<9% or >=9%), and concomitant SU use at screening as factors, and baseline value of the fasting plasma glucose as a covariate. Null hypothesis: no difference between treatments in change from baseline fasting plasma glucose. Power: based on the primary measurement; Test type: Superiority or Other; p < .0001, ANCOVA; Least Squares Mean Difference = -16.9, 95% CI 2-sided [-24.4 to -9.4], Standard Error of Mean 3.80

15. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline to Week 364
Description: Change in fasting plasma glucose from baseline (Day -3) to Week 364.
Time Frame: Day -3, Week 364
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Exenatide Once Weekly -> Exenatide Once Weekly | Exenatide Twice Daily -> Exenatide Once Weekly | All Treatment
Number analyzed (Participants) | 58 | 64 | 122
mg/dL | -18.3 (2.97) [-30.8 to -5.7] | -27.7 (2.90) [-39.0 to -16.4] | -23.6 [-33.0 to -14.2]

16. Secondary Outcome: Change in Blood Pressure From Baseline to Week 30
Description: Change in Sitting Diastolic Blood Pressure and Sitting Systolic Blood Pressure from baseline to Week 30
Time Frame: Day -3, Week 30
Population: ITT Population using observed data.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 126 | 130
mmHg
  Sitting Systolic Blood Pressure | -4.4 (1.04) | -3.8 (1.28)
  Sitting Diastolic Blood Pressure | -1.1 (0.76) | -2.3 (0.83)

17. Secondary Outcome: Change in Blood Pressure From Baseline to Week 364
Description: Change in Sitting Diastolic Blood Pressure and Sitting Systolic Blood Pressure from baseline to Week 364
Time Frame: Day -3, Week 364
Population: 7-Year Completer Population using observed data.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Exenatide Twice Daily -> Exenatide Once WeeklyEdit: Subcutaneous injection of exenatide, twice a day (5 mcg exenatide per dose for first 4 weeks, then 10 mcg exenatide per dose for 26 weeks) followed by 2 mg exenatide, once a week.
Arm/Group | Exenatide Once Weekly -> Exenatide Once Weekly | Exenatide Twice Daily -> Exenatide Once WeeklyEdit | All Treatment
Number analyzed (Participants) | 58 | 64 | 122
mmHg
  Sitting Systolic Blood Pressure | 1.3 (16.21) | 1.0 (17.32) | 1.2 (16.73)
  Sitting Diastolic Blood Pressure | -1.7 (8.87) | -3.6 (9.59) | -2.7 (9.26)

18. Secondary Outcome: Change in Total Cholesterol From Baseline to Week 30
Description: Change in total cholesterol from baseline (Day -3) to Week 30.
Time Frame: Day -3, Week 30
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 139 | 137
mg/dL | -11.9 (2.29) [-16.4 to -7.4] | -3.8 (2.35) [-8.4 to 0.8]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Analysis: Change in total cholesterol from baseline (Day -3) to Week 30 was analyzed using an ANCOVA model including treatment, baseline HbA1c stratum (<9% or >=9%), and concomitant SU use at screening as factors, and baseline value of the total cholesterol as a covariate. Null hypothesis: no difference between treatments in change from baseline total cholesterol. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.0077, ANCOVA; Least Squares Mean Difference = -8.2, 95% CI 2-sided [-14.1 to -2.2], Standard Error of Mean 3.04

19. Secondary Outcome: Change in Total Cholesterol From Baseline to Week 364
Description: Change in total cholesterol from baseline (Day -3) to Week 364.
Time Frame: Day -3, Week 364
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Exenatide Once Weekly -> Exenatide Once Weekly | Exenatide Twice Daily -> Exenatide Once Weekly | All Treatment
Number analyzed (Participants) | 58 | 64 | 122
mg/dL | -15.0 (2.29) [-23.6 to -6.4] | -4.8 (2.35) [-13.0 to 3.3] | -9.6 [-16.2 to -3.0]

20. Secondary Outcome: Change in High-density Lipoprotein Cholesterol (HDL-C) From Baseline to Week 30
Description: Change in high-density lipoprotein cholesterol (HDL-C) from baseline (Day -3) to Week 30.
Time Frame: Day -3, Week 30
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 139 | 137
mg/dL | -0.9 (0.56) [-2.0 to 0.2] | -1.3 (0.57) [-2.5 to -0.2]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Analysis: Change in HDL-C from baseline (Day -3) to Week 30 was analyzed using an ANCOVA model including treatment, baseline HbA1c stratum (<9% or >=9%), and concomitant SU use at screening as factors, and baseline value of the HDL as a covariate. Null hypothesis: no difference between treatments in change from baseline HDL. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.5613, ANCOVA; Least Squares Mean Difference = 0.4, 95% CI 2-sided [-1.0 to 1.9], Standard Error of Mean 0.74

21. Secondary Outcome: Change in High-density Lipoprotein Cholesterol (HDL-C) From Baseline to Week 364
Description: Change in high-density lipoprotein cholesterol (HDL-C) from baseline (Day -3) to Week 364.
Time Frame: Day -3, Week 364
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Exenatide Once Weekly -> Exenatide Once Weekly | Exenatide Twice Daily -> Exenatide Once Weekly | All Treatment
Number analyzed (Participants) | 58 | 64 | 122
mg/dL | 2.2 (0.56) [-0.2 to 4.7] | 3.4 (0.57) [1.0 to 5.7] | 2.8 [1.0 to 4.7]

22. Secondary Outcome: Change in Low-density Lipoprotein Cholesterol (LDL-C) From Baseline to Week 364
Description: Change in low-density lipoprotein cholesterol (LDL-C) from baseline (Day -3) to Week 364.
Time Frame: Day -3, Week 364
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Exenatide Once Weekly -> Exenatide Once Weekly | Exenatide Twice Daily -> Exenatide Once Weekly | All Treatment
Number analyzed (Participants) | 58 | 64 | 122
mg/dL | -13.6 (0.56) [-21.3 to -6.0] | -7.5 (0.57) [-14.7 to -0.3] | -10.4 [-16.2 to -4.6]

23. Secondary Outcome: Ratio of Triglycerides at Week 30 to Baseline
Description: Ratio of triglycerides (measured in mg/dL) at Week 30 to baseline (Day -3). Log (Postbaseline Triglycerides) - log (Baseline Triglycerides); change from baseline to endpoint is presented as ratio of endpoint to baseline.
Time Frame: Day -3, Week 30
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exenatide Once Weekly | Exenatide Twice Daily
Number analyzed (Participants) | 139 | 137
ratio | 0.85 (0.029) [0.80 to 0.91] | 0.89 (0.031) [0.84 to 0.96]
Statistical Analysis 1: Comparison: Exenatide Once Weekly vs Exenatide Twice Daily; Analysis: Triglycerides data were logarithm-transformed and the change at Week 30 to baseline (Day -3), expressed as the ratio, was analyzed by an ANCOVA model including treatment, baseline HbA1c stratum (<9% or >=9%), and concomitant SU use at screening as factors, and baseline value of the triglycerides as a covariate. Null hypothesis: no difference between treatments in change from baseline triglycerides. Power: based on the primary measurement; Test type: Superiority or Other; p = 0.2915, ANCOVA; Geometic Least Squares Mean Ratio = 0.95, 95% CI 2-sided [0.87 to 1.04], Standard Error of Mean 0.042

24. Secondary Outcome: Ratio of Triglycerides at Week 364 to Baseline
Description: Ratio of triglycerides (measured in mg/dL) at Week 364 to baseline (Day -3). Log (Postbaseline Triglycerides) - log (Baseline Triglycerides); change from baseline to endpoint is presented as ratio of endpoint to baseline.
Time Frame: Day -3, Week 364
Population: as for outcome 13
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Exenatide Once Weekly -> Exenatide Once Weekly | Exenatide Twice Daily -> Exenatide Once Weekly | All Treatment
Number analyzed (Participants) | 58 | 64 | 122
ratio | 0.91 (0.029) [0.80 to 1.02] | 0.94 (0.031) [0.84 to 1.06] | 0.93 [0.85 to 1.01]

25. Secondary Outcome: Assessment on Event Rate of Treatment-emergent Hypoglycemic Events With SU Use at Screening
Description: The major hypoglycemia category included events that, in the judgment of the investigator or physician, resulted in loss of consciousness, seizure, coma, or other change in mental status consistent with neuroglycopenia, in which symptoms resolved after administration of intramuscular glucagon or intravenous glucose, required third-party assistance, and was accompanied by a blood glucose concentration of less than 54 mg/dL prior to treatment, whether or not symptoms of hypoglycemia were perceived by the subject. The minor hypoglycemia were accompanied by a blood glucose concentration of less than 54 mg/dL prior to treatment and not classified as major hypoglycemia.
Time Frame: Day 1 to Week 364
Population: ITT Population who participated in the 30-week assessment period and using SU at screening.
Measure: Mean (Standard Error); unit: events per subject-year
Groups:
- Exenatide Once Weekly With SU: Subjects subcutaneous injection of 2 mg exenatide, once a week using concomitant SU at screening. Week 0 to week 30.
- Exenatide Twice Daily With SU: Subjects with subcutaneous injection of exenatide, twice a day (5 mcg exenatide per dose for first 4 weeks, then 10 mcg exenatide per dose for 26 weeks) using concomitant SU at screening. Week 0 to week 30.
- Exenatide Once Weekly -> Exenatide Once Weekly With SU: Subjects subcutaneous injection of 2 mg exenatide, once a week using concomitant SU at screening. Week 31 to week 364
- Exenatide Twice Daily -> Exenatide Once Weekly With SU: Subjects with subcutaneous injection of exenatide, twice a day (5 mcg exenatide per dose for first 4 weeks, then 10 mcg exenatide per dose for 26 weeks) followed by 2 mg exenatide, once a week using concomitant SU at screening. Week 31 to week 364.
- Exenatide Once Weekly With SU: Subcutaneous injection of 2 mg exenatide, once a week using concomitant SU at screening. Pooling unique subjects from exenatide once weekly (WK 0-30), exenatide once weekly -> exenatide once weekly (WK 31-364), and exenatide twice daily -> exenatide once weekly (WK 31-364).
Arm/Group | Exenatide Once Weekly With SU | Exenatide Twice Daily With SU | Exenatide Once Weekly -> Exenatide Once Weekly With SU | Exenatide Twice Daily -> Exenatide Once Weekly With SU | Exenatide Once Weekly With SU
Number analyzed (Participants) | 55 | 52 | 49 | 50 | 105
events per subject-year
  Major hypoglycemic events | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Minor hypoglycemic events | 0.57 (0.139) | 0.38 (0.113) | 0.49 (0.046) | 0.22 (0.029) | 0.36 (0.026)

26. Secondary Outcome: Assessment on Event Rate of Treatment-emergent Hypoglycemic Events With Non-SU Use at Screening
Description: as for outcome 25
Time Frame: Day 1 to Week 364
Population: ITT Population who participated in the 30-week assessment period and not using SU at screening.
Measure: Mean (Standard Error); unit: events per subject-year
Groups:
- Exenatide Once Weekly With Non-SU: Subjects subcutaneous injection of 2 mg exenatide, once a week not using concomitant SU at screening. Week 0 to week 30.
- Exenatide Twice Daily With Non-SU: Subjects with subcutaneous injection of exenatide, twice a day (5 mcg exenatide per dose for first 4 weeks, then 10 mcg exenatide per dose for 26 weeks) not using concomitant SU at screening. Week 0 to week 30.
- Exenatide Once Weekly -> Exenatide Once Weekly With Non-SU: Subjects subcutaneous injection of 2 mg exenatide, once a week not using concomitant SU at screening. Week 31 to week 364
- Exenatide Twice Daily -> Exenatide Once Weekly With Non-SU: Subjects with subcutaneous injection of exenatide, twice a day (5 mcg exenatide per dose for first 4 weeks, then 10 mcg exenatide per dose for 26 weeks) followed by 2 mg exenatide, once a week not using concomitant SU at screening. Week 31 to week 364.
- Exenatide Once Weekly With Non-SU: Subcutaneous injection of 2 mg exenatide, once a week not using concomitant SU at screening. Pooling unique subjects from exenatide once weekly (WK 0-30), exenatide once weekly -> exenatide once weekly (WK 31-364), and exenatide twice daily -> exenatide once weekly (WK 31-364).
Arm/Group | Exenatide Once Weekly With Non-SU | Exenatide Twice Daily With Non-SU | Exenatide Once Weekly -> Exenatide Once Weekly With Non-SU | Exenatide Twice Daily -> Exenatide Once Weekly With Non-SU | Exenatide Once Weekly With Non-SU
Number analyzed (Participants) | 93 | 93 | 79 | 80 | 173
events per subject-year
  Major hypoglycemic events | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.000)
  Minor hypoglycemic events | 0.00 (0.000) | 0.02 (0.020) | 0.03 (0.009) | 0.06 (0.013) | 0.04 (0.007)

ADVERSE EVENTS:
Groups:
- Exenatide Once Weekly (WK 0-30); Exenatide Once Weekly -> Exenatide Once Weekly (WK 31-364): Subcutaneous injection of 2 mg exenatide, once a week.
- Exenatide Twice Daily (WK 0-30): Subcutaneous injection of exenatide, twice a day (5 mcg exenatide per dose for first 4 weeks, then 10 mcg exenatide per dose for 26 weeks).
- Exenatide Twice Daily -> Exenatide Once Weekly (WK 31-364): Subcutaneous injection of exenatide, twice a day (5 mcg exenatide per dose for first 4 weeks, then 10 mcg exenatide per dose for 26 weeks) followed by 2 mg exenatide, once a week.
- Exenatide Once Weekly: Subcutaneous injection of 2 mg exenatide, once a week. Pooling unique subjects from exenatide once weekly (WK 0-30), exenatide once weekly -> exenatide once weekly (WK 31-364), and exenatide twice daily -> exenatide once weekly (WK 31-364).
Arm/Group | Exenatide Once Weekly (WK 0-30) | Exenatide Twice Daily (WK 0-30) | Exenatide Once Weekly -> Exenatide Once Weekly (WK 31-364) | Exenatide Twice Daily -> Exenatide Once Weekly (WK 31-364) | Exenatide Once Weekly
Serious Adverse Events (participants affected / at risk) | 8/148 | 5/145 | 36/128 | 29/130 | 71/278
Other Adverse Events (participants affected / at risk) | 124/148 | 106/145 | 121/128 | 122/130 | 265/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (WK 0-30) (N=148) | Exenatide Twice Daily (WK 0-30) (N=145) | Exenatide Once Weekly -> Exenatide Once Weekly (WK 31-364) (N=128) | Exenatide Twice Daily -> Exenatide Once Weekly (WK 31-364) (N=130) | Exenatide Once Weekly (N=278)
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 1 | 3
Cerebral artery occlusion (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 2
Diverticulitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 3
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 1 | 3
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Tooth impacted (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 2
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 2 | 6
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 3 | 0 | 3
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 2 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2 | 1 | 3
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 2 | 1 | 3
Coronary artery disease (Cardiac disorders) | 0 | 0 | 4 | 0 | 4
Coronary artery occlusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Macular oedema (Eye disorders) | 0 | 0 | 1 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 2 | 2
Device dislocation (General disorders) | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 2 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 3 | 0 | 3
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 2
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Herpes zoster oticus (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Infected bites (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Perirectal abscess (Infections and infestations) | 0 | 0 | 1 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 2
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hyperlactacidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 2
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 2
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (WK 0-30) (N=148) | Exenatide Twice Daily (WK 0-30) (N=145) | Exenatide Once Weekly -> Exenatide Once Weekly (WK 31-364) (N=128) | Exenatide Twice Daily -> Exenatide Once Weekly (WK 31-364) (N=130) | Exenatide Once Weekly (N=278)
Nausea (Gastrointestinal disorders) | 40 | 49 | 26 | 25 | 82
Injection site pruritus (General disorders) | 27 | 2 | 5 | 9 | 40
Diarrhoea (Gastrointestinal disorders) | 24 | 18 | 35 | 34 | 79
Constipation (Gastrointestinal disorders) | 15 | 9 | 11 | 16 | 40
Vomiting (Gastrointestinal disorders) | 16 | 27 | 21 | 21 | 54
Urinary tract infection (Infections and infestations) | 15 | 11 | 23 | 30 | 63
Gastroenteritis viral (Infections and infestations) | 12 | 8 | 18 | 11 | 37
Upper respiratory tract infection (Infections and infestations) | 12 | 25 | 54 | 64 | 124
Dyspepsia (Gastrointestinal disorders) | 11 | 3 | 7 | 9 | 26
Injection site erythema (General disorders) | 11 | 0 | 7 | 6 | 21
Fatigue (General disorders) | 9 | 5 | 11 | 12 | 31
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 | 6 | 15 | 13 | 39
Nasopharyngitis (Infections and infestations) | 10 | 8 | 34 | 41 | 78
Headache (Nervous system disorders) | 9 | 7 | 15 | 15 | 38
Injection site bruising (General disorders) | 7 | 14 | 7 | 10 | 24
Sinusitis (Infections and infestations) | 7 | 10 | 26 | 35 | 66
Dizziness (Nervous system disorders) | 5 | 9 | 10 | 10 | 25
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 8 | 5 | 15
Cataract (Eye disorders) | 2 | 0 | 15 | 9 | 25
Abdominal discomfort (Gastrointestinal disorders) | 5 | 2 | 8 | 8 | 19
Abdominal pain (Gastrointestinal disorders) | 5 | 3 | 8 | 8 | 20
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 7 | 8 | 17
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 11 | 10 | 22
Toothache (Gastrointestinal disorders) | 1 | 3 | 6 | 9 | 16
Seasonal allergy (Immune system disorders) | 2 | 2 | 13 | 5 | 20
Bronchitis (Infections and infestations) | 4 | 6 | 18 | 25 | 46
Conjunctivitis (Infections and infestations) | 1 | 2 | 6 | 9 | 16
Ear infection (Infections and infestations) | 0 | 1 | 6 | 7 | 13
Gastroenteritis (Infections and infestations) | 0 | 0 | 9 | 6 | 15
Herpes zoster (Infections and infestations) | 1 | 1 | 7 | 10 | 18
Influenza (Infections and infestations) | 2 | 3 | 11 | 17 | 30
Onychomycosis (Infections and infestations) | 0 | 0 | 6 | 7 | 13
Tooth abscess (Infections and infestations) | 3 | 1 | 7 | 7 | 17
Tooth infection (Infections and infestations) | 4 | 1 | 10 | 7 | 20
Contusion (Injury, poisoning and procedural complications) | 3 | 1 | 12 | 10 | 25
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 12 | 10 | 24
Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 6 | 8 | 14
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 3 | 6 | 10 | 17
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 13 | 8 | 21
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 7 | 6 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 6 | 25 | 28 | 58
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 7 | 10 | 19
Oedema peripheral (General disorders) | 1 | 0 | 6 | 14 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 6 | 27 | 25 | 55
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 5 | 10 | 16
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 3 | 12 | 13 | 28
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 23 | 15 | 40
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 2 | 4 | 11 | 19
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 15 | 10 | 26
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 21 | 22 | 44
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5 | 8 | 13
Anxiety (Psychiatric disorders) | 2 | 3 | 10 | 6 | 18
Depression (Psychiatric disorders) | 2 | 4 | 10 | 12 | 24
Insomnia (Psychiatric disorders) | 4 | 4 | 9 | 11 | 24
Nephrolithiasis (Renal and urinary disorders) | 2 | 1 | 13 | 9 | 23
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 7 | 6 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 14 | 14 | 33
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 8 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 8 | 12 | 21
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 7 | 9 | 16
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 14 | 8 | 22
Hypertension (Vascular disorders) | 5 | 4 | 22 | 22 | 49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less